CLINICAL TRIAL: NCT00719693
Title: Assessment of the Effect of Food on ABT-143 Bioavailability
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M10-442
Record Dates: First submitted 2008-07-18; First posted 2008-07-22 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Pharmacokinetic Variables
Keywords: Food effect, phase I; adverse events
MeSH Terms: interventions — Rosuvastatin Calcium; fenofibric acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): ABT-143 under low-fat meal condition
  Interventions: Drug: ABT-143 ( rosuvastatin calcium and fenofibric acid )
- B (Experimental): ABT-143 under fasting meal condition
  Interventions: Drug: ABT-143 (rosuvastatin calcium and fenofibric acid )

INTERVENTIONS:
Drug: ABT-143 ( rosuvastatin calcium and fenofibric acid ) — one dose under low-fat meal condition
  Other Names: ABT-143; fenofibric acid/rosuvastatin calcium
  Arms: A
Drug: ABT-143 (rosuvastatin calcium and fenofibric acid ) — one dose under fasting meal condition
  Arms: B

SUMMARY:
Single-dose, open-label, two-period crossover study of ABT-143

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years of age (inclusive)
* BMI 19 to 29 inclusive

Exclusion Criteria:

* Asian ancestry
* Concurrent participation in another study
* Females pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | 7 days

SECONDARY OUTCOMES:
Adverse Events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (1):
- Site Reference ID/Investigator# 9242, Evansville, Indiana, United States